CLINICAL TRIAL: NCT04427423
Title: Experimental-controlled, Randomized, Single Blind Trial of Effectiveness of Positional Distraction With Stabilization Exercises Versus Stabilization Exercises Alone in the Management of Lumbar Radiculopathy.
Brief Title: Positional Distraction and Stabilization Exercises in Adults With Lumbar Radiculopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SKhan
Record Dates: First submitted 2020-04-27; First posted 2020-06-11 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: All the patients will be randomly allocated into treatment and control groups 50 in experimental and 50 in control group. The treatment group will receive positional with stabilization exercises while the control group will be treated with stabilization exercises only.
Who Masked: Participant
Masking Description: The patients were blinded from the treatment groups that either he/she are in experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional Distraction plus Stabilization Exercise group (Experimental): The treatment group will receive positional distraction with stabilization exercises
  Interventions: Other: physical therapy treatment
- Stabilization Exercise group (Active Comparator): control group will be treated with stabilization exercises only.
  Interventions: Other: physical therapy treatment

INTERVENTIONS:
Other: physical therapy treatment — the experimental group received positional distraction plus stabilization exercises and the control group received stabilization exercises only.

SUMMARY:
This study evaluate the addition of positional distraction to stabilization exercises in the treatment of lumbar radiculopathy in adults. Half of the patients will recieve positional distraction and stabilization exercises in combination, while the other half will recieve stabilization exercises only.

DETAILED DESCRIPTION:
In positioanl distraction making use of the body position to produce traction at an isolated spinal level to maximally open the affected neuroforamen. It is an alternative to lumbar mechanical traction.

The spinal level of vertebral level requiring traction is palpated and a soft roll is placed and the patient side lies on the unaffected side. For further distraction both hips are flexed until movement is noted at the spinal level needing traction.

Further, distraction applied by rotating upper trunk to opposite side of pain.

Stabilization exercises are mainly used for the stability of joints and for improving muscle strength.

The first step of lumbar stabilization exercises are to maintain functional back positions during all activities. The second step is to improve strength and endurance of the core muscles.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lumbar radiculopathy
* Age limit 30-50 years
* Both males and females
* Pain history more than 12 weeks but less than one year
* Patient having lumbar disc bulge at maximum two adjacent levels

Exclusion Criteria:

* Any type of tumor and infection in the spine
* Spondylolisthesis at L4- L5, L5-S1
* Fracture of the lumbar spine
* Sciatica other than lumbar region (piriformis syndrome)
* Acute cardiopulmonary conditions
* Morbid obesity (BMI > 30)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain intensity at 8 weeks | All the subjects were assessed before and after 8 weeks of treatment.
  The pain intensity measured on self reported Visual Analogue Scale. (0 means no pain and 10 is the high intensity of pain).
Change from baseline Disability at 8 weeks | All the subjects were assessed before and after 8 weeks of treatment.
  The disability were assessed on Roland Morris Disability Questionnaire. where 0 means no disability and 24 is the high disability.

CONTACTS AND LOCATIONS:
Overall Officials: IPMR DUHS, Study Director — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan S, Hasnain F, Soomro RR, Rehmani A. Comparison of positional distraction with stabilisation exercises versus stabilisation exercises alone in the management of lumbar radiculopathy: A randomized controlled-trial. J Pak Med Assoc. 2024 Jan;74(1):5-9. doi: 10.47391/JPMA.6540. PMID 38219156